CLINICAL TRIAL: NCT02161211
Title: Dismantling the Components and Dosing of CBT for Co-Occurring Disorders
Acronym: CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSYCH-2016-22016
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-05

CONDITIONS: CBT Decoupling; CBT Anxiety Reduction; CBT Combined
Keywords: alcohol; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- De-coupling (Experimental): Six sessions of CBT for anxiety-alcohol de-coupling
  Interventions: Behavioral: De-coupling
- Anxiety Reduction (Experimental): Six sessions of CBT for anxiety reduction.
  Interventions: Behavioral: Anxiety Reduction
- Combined (Experimental): Three sessions devoted to anxiety reduction and to anxiety-alcohol de-coupling each.
  Interventions: Behavioral: Combined

INTERVENTIONS:
Behavioral: De-coupling — Six sessions of CBT for anxiety-alcohol de-coupling
  Arms: De-coupling
Behavioral: Anxiety Reduction — Six sessions of CBT for anxiety reduction.
  Arms: Anxiety Reduction
Behavioral: Combined — Three sessions devoted to anxiety reduction and to anxiety-alcohol de-coupling each.
  Arms: Combined

SUMMARY:
The purpose of this study is to establish a brief CBT intervention that can largely, if not fully eliminate the deleterious effect of common co-occurring anxiety disorders on alcohol use disorder treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic and Statistical Manual IV diagnosis of panic disorder, generalized anxiety disorder, and/or social anxiety disorder within the past 30 days;
* inpatient treatment at Lodging Plus primarily for alcohol (vs. other drug) dependence
* alcohol use in the 30 days preceding the study
* ability to provide informed consent
* minimum of a sixth grade reading level (deemed necessary to complete study materials);
* willingness to provide contact information to confirm study follow-up appointments
* lives within proximity to the Twin Cities (e.g., within about an hour's drive) for the purpose attending follow-up visits

Exclusion Criteria:

* lifetime history of psychosis or mania by history
* cognitive or physical impairment that precludes study participation
* currently and seriously suicidal (i.e., plan and intent)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Kushner, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Lodging Plus Program, Fairview Hospital, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | De-coupling | Anxiety Reduction | Combined
Started | 92 | 94 | 93
Completed | 59 | 62 | 63
Not Completed | 33 | 32 | 30
Not completed — Lost to Follow-up | 21 | 27 | 21
Not completed — Dropped | 12 | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | De-coupling | Anxiety Reduction | Combined | Total
Number analyzed (Participants) | 92 | 94 | 93 | 279
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38.5 [31 to 49] | 43 [33 to 51] | 38 [32 to 49] | 40 [32 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 36 | 35 | 105
  Male | 58 | 58 | 58 | 174
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 6 | 11
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 8 | 17
  White | 82 | 81 | 71 | 234
  More than one race | 1 | 6 | 8 | 15
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 92 | 94 | 93 | 279

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Relapsed to Drinking at 4 Months
Description: Relapse status will be assessed using categorical relapse status (yes vs. no). Count is of those who relapsed
Time Frame: 4 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | De-coupling | Anxiety Reduction | Combined
Number analyzed (Participants) | 63 | 78 | 67
Participants | 30 | 43 | 35
Statistical Analysis 1: Comparison: De-coupling vs Anxiety Reduction vs Combined; Null hypothesis = no difference in frequency in relapse between groups; Test type: Superiority; p = .673, Chi-squared; df = 2

2. Primary Outcome: Number of Drinking Days in 4 Months Post Treatment
Description: Negative binomial regression with offset for possible drinking days exposure in 4 months post treatment
Time Frame: 4-months
Measure: Mean (Standard Error); unit: drinking days
Arm/Group | De-coupling | Anxiety Reduction | Combined
Number analyzed (Participants) | 63 | 78 | 67
drinking days | 8.44 (1.13) | 13.04 (1.53) | 11.34 (1.45)
Statistical Analysis 1: Comparison: De-coupling vs Combined; Test type: Superiority; p = .133, Wald Chi-squared; Negative binomial regression with offset of natural log of possible drinking days; Wald Chi-squared = -.278, 95% CI 2-sided [-.64 to .084]
Statistical Analysis 2: Comparison: Anxiety Reduction vs Combined; Test type: Superiority; p = .562, Wald Chi-squared; Wald Chi-squared = .101, 95% CI 2-sided [-.24 to .44]

3. Primary Outcome: Number of Standard Drinks Per Drinking Day
Description: Drinks per drinking day among those who relapsed by 4 months. Standard Drink is defined as 12oz beer, 4ox wine, 3oz fortified wine, 1oz hard liquor
Time Frame: 4 months
Measure: Mean (Standard Error); unit: drinks per drinking day
Arm/Group | De-coupling | Anxiety Reduction | Combined
Number analyzed (Participants) | 30 | 43 | 35
drinks per drinking day | 17.17 (2.50) | 17.72 (2.08) | 17.67 (2.31)
Statistical Analysis 1: Comparison: De-coupling vs Combined; Test type: Superiority; p = .982, ANOVA; F(2,105) = .019

4. Secondary Outcome: Number of Participants Who Met SCID-IV Criteria for Alcohol Dependence at 4 Months
Description: Relapse to Diagnostic and Statistical Manual (DSM)-IV alcohol dependence criteria based on Structured Clinical Interview for DSM-IV (SCID) at 4 months
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | De-coupling | Anxiety Reduction | Combined
Number analyzed (Participants) | 63 | 78 | 67
Participants | 13 | 21 | 16
Statistical Analysis 1: Comparison: De-coupling vs Anxiety Reduction vs Combined; Null hypothesis = no difference in proportion between the groups; Test type: Superiority; p = .685, Chi-squared

5. Secondary Outcome: Number of Participants Who Relapsed to Hazardous Drinking
Description: Relapse to hazardous drinking (hazardous drinking is defined as 3 or more per occasion for women or more than 7 drinks per week, 4 or more per occasion for men or more than 14 drinks per week) at 4 months
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | De-coupling | Anxiety Reduction | Combined
Number analyzed (Participants) | 63 | 78 | 67
Participants | 27 | 39 | 34
Statistical Analysis 1: Comparison: De-coupling vs Anxiety Reduction vs Combined; Null hypothesis = no significant difference in frequency of hazardous drinking between groups; Test type: Superiority; p = .608, Chi-squared

ADVERSE EVENTS:
Time Frame: Through 8 month follow-up
Arm/Group | De-coupling | Anxiety Reduction | Combined
All-Cause Mortality (participants affected / at risk) | 0/92 | 1/94 | 1/93
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/94 | 0/93
Other Adverse Events (participants affected / at risk) | 0/92 | 0/94 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02161211/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT02161211/ICF_000.pdf